CLINICAL TRIAL: NCT03056014
Title: Supplementation of N-acetylcysteine and Arachonic Acid in Type 1 Diabetes to Determine Changes in Oxidative Stress
Brief Title: Antioxidant Use in Diabetes to Reduce Oxidative Stress
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Sarah Crimmins, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00067782
Record Dates: First submitted 2017-01-30; First posted 2017-02-16 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Ameliorating Oxidative Stress in Type 1 Diabetes
MeSH Terms: interventions — Acetylcysteine; Fatty Acids, Unsaturated

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- N-acetylcysteine 600 mg (Active Comparator)
  Interventions: Drug: N-acetyl cysteine
- N-acetylcysteine 1200 mg (Active Comparator)
  Interventions: Drug: N-acetyl cysteine
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- PUFA 1000 mg (Active Comparator)
  Interventions: Dietary Supplement: omega 6 Fish oil ( PUFA)
- PUFA 2000 mg (Active Comparator)
  Interventions: Dietary Supplement: omega 6 Fish oil ( PUFA)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — giving varying doses of NAC in order to determine which reduces oxidative stress.
  Arms: N-acetylcysteine 1200 mg; N-acetylcysteine 600 mg
Dietary Supplement: omega 6 Fish oil ( PUFA) — giving varying doses of PUFA in order to determine which reduces oxidative stress.
  Arms: PUFA 1000 mg; PUFA 2000 mg
Dietary Supplement: Placebo — L-alanine placebo pill to determine if effect is supplement related or random effect.
  Arms: Placebo; placebo

SUMMARY:
Dietary supplementation with antioxidant vitamins, such as Vitamin C and Vitamin E, reduces malformation rates in embryos of diabetic animals. However, human trials exploring the benefits of these antioxidant vitamins have produced unsatisfactory results in trials designed to alleviating diabetic retinopathy, cardiovascular disease, and preeclampsia in pregnancies. The investigators hypothesize that more potent, and better-targeted antioxidants, such as N-acetylcysteine (NAC) and Polyunsaturated Fatty Acids(PUFA), will be successful in preventing birth defects in the offspring of women with diabetes.

DETAILED DESCRIPTION:
Specific Aim 1. Recruit non pregnant women with T1DM and investigate the efficacy of dietary NAC on ameliorating oxidative stress Study design. Diabetic patients will be provided with NAC or placebo for 14 days, while receiving usual clinical care. The oxidative stress status will be assessed by measuring biomarkers in blood samples pre and post intervention. In addition to a placebo control group, three treatment groups including Group 1 (NAC 600 mg/day), Group 2 (NAC 1200 mg/day), and Group 3 (NAC 1800 mg/day) will be studied. The choice of dosage of NAC is based on published studies, which show effectiveness of NAC in 600 or 1200 mg day in alleviating oxidative stress in diabetic patients, both in men and women, without adverse side effects. The investigators will use the supplement company TwinLab for our study. The university of Maryland Pharmacy department will analyze the NAC for purity prior to starting the study. At day 7, participants will be called via phone assess for symptoms and side effects from medications. All participants will be called. At the end of 14 days, the patients will return to the CDE with a survey asking about compliance with medication and any side effects. They will also bring the pill bottle so that study personnel can do a pill count. At this time blood will be draw for the biomarker levels to look for changes in oxidative stress.

Specific Aim 2. To investigate effect of PUFAs on ameliorating oxidative stress in diabetic non-pregnant women.

Study design: The investigators will recruit a new group of Non-pregnant women with T1DM will be enrolled and randomly assigned to placebo or one of three treatment groups. Study volunteers will be divided into 1 of 3 groups. PUFA; Group 1 (1000 mg/day) or Group 2 (2000 mg/day) or Group 3(placebo). The treatment regimens, sample collection, biomarker assessment, side effect monitoring and statistical analysis will be performed as described in SA 1. The investigators will perform an analysis of the oxidative stress biomarkers as described in SA1. The investigators will use TwinLab as our commercial supplier of PUFA for our trial. There fish oil supplements have been involved in greater than 40 published trials. The fish oil supplement will be analyzed by the University of Maryland pharmacy department prior to starting the study to analyze for purity.

Specific Aim 3: To investigate the potential secondary benefit of NAC/PUFA on kidney function and lipid profile. Urine and serum samples will be collected on all enrolled subjects at day 0 and Day 14 to monitor for improvement in microalbumin in the urine and lipid profile in the serum. Previous studies have shown improvements in LDL with supplementation of NAC. The investigators will look at how various dosages effect the improvement in microalbumin and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* hemoglobin a1c <10
* type 1 diabetes

Exclusion Criteria:

* pregnancy
* BMI > 40
* greater than 1 alcoholic beverages per week
* any tobacco use
* prescribed nitroglycerin, HIV protease inhibits, corticosteroids, cephalosporins, or blood thinners
* vascular complications(history of coronary artery disease, cerebral vascular accident, transient ischemic attack, claudication).

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — we specifically want to study this in reproductive age females.
Enrollment: 8 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in level of oxidative stress with varying doses of NAC at 2 weeks. | 2 weeks
Change from baseline in level of oxidative stress with varying doses of omega 6 fish oil(PUFA) at 2 weeks. | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No